CLINICAL TRIAL: NCT01069393
Title: Improving Management of Type 1 Diabetes in the UK: The DAFNE Programme as a Research Test-bed - 5 x 1 Day RCT
Brief Title: Alternative Delivery of Dose Adjustment For Normal Eating (DAFNE) Trial in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University Hospitals, Leicester (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); Northumbria Healthcare NHS Foundation Trust (Other); NHS Greater Glasgow and Clyde (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH15581
Record Dates: First submitted 2010-02-10; First posted 2010-02-17 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard DAFNE (Active Comparator): Usual DAFNE course taught over 5 consecutive days in one week
  Interventions: Other: DAFNE course (Timing of delivery of education)
- DAFNE 5x1 day (Experimental): DAFNE course taught 1 day a week for 5 consecutive weeks
  Interventions: Other: DAFNE course (Timing of delivery of education)

INTERVENTIONS:
Other: DAFNE course (Timing of delivery of education) — Education delivered over one day a week for 5 consecutive weeks, as opposed to 5 consecutive days over 1 week.

SUMMARY:
The best format for the delivery of structured education for adults with Type 1 diabetes is unclear. Currently some hospitals invite their patients to attend a 5 day outpatient course run over one week (Dose Adjustment For Normal Eating (DAFNE)). Other centres offer 1 day a week for 3 to 5 weeks. We aim to find out whether or not the benefit of benefits are the same then it would mean that the course could routinely be offered to patients in either format, thus allowing more patient choice and flexibility.

DETAILED DESCRIPTION:
The DAFNE (Dose Adjustment for Normal Eating) course is a 1-week structured education course teaching skills in insulin use and dietary freedom to individuals with Type 1 diabetes. At the moment, we do not understand enough about why some people get more out of the DAFNE programmes than others. Currently DAFNE is always taught over 1 week. We aim to find out whether or not the benefit of DAFNE is the same whether it is delivered over 5 consecutive days, or one day a week for 5 consecutive weeks. If the benefits are the same then it would mean that the course could routinely be offered to patients in either format, thus allowing more patient choice and flexibility. At present there have been no RCTs to address

Approximately 170 people will take part in this study over the next 2 years. Half the people who participate will be allocated to attend a DAFNE course over 5 consecutive days, and the other halfwill attend one day a week for 5 consecutive weeks. We will perform routine biomedical assessments as part of the DAFNE programme and normal diabetes care (e.g. HbA1c (a measure of long-term blood glucose control), weight, blood pressure, blood biochemistry), and ask patients to recall hypoglycaemic (low blood sugar) events. We will also ask participants to fill in some research questionnaires, they will take 45-60 minutes to fill in each time. They will include questions about their diabetes, quality of life, well-being and diabetes knowledge. These assessments will be made at 3 time points; baseline, 6 and 12 months.

The main outcome measure is change in HbA1c, with the other biomedical and psychosocial parameters being of secondary importance. These evaluations will help us develop the DAFNE programme further and inform us how best to deliver the course in the future.

ELIGIBILITY:
Inclusion Criteria:

* adults with Type 1 diabetes for at least 6 months
* HbA1c <12%
* willing to undertake intensive insulin therapy

Exclusion Criteria:

* severe diabetic complications (making group education difficult)
* inability to communicate in English
* strong preference for on attending a one week course or one day a week for 5 consecutive weeks
* inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Improvement in HbA1c (glycosylated haemoglobin) | 6 & 12 months

SECONDARY OUTCOMES:
Number of severe hypoglycaemic episodes | 12 months
Psychosocial measures, such as quality of life, emotional well-being, self-efficacy,will be assessed via questionnaires | 12 months
Qualitative evaluation via in-depth interviews to assess patients' experiences of the intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon Heller, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Greater Glasgow & Clyde, Glasgow
  - East Lancashire Hospitals NHS Trust, Lancashire
  - University Hospitals, Leicester, Leicester
  - University College London, London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norfolk
  - Northumbria Healthcare NHS Foundation Trust, Northumbria

REFERENCES:
- [Derived] Elliott J, Lawton J, Rankin D, Emery C, Campbell M, Dixon S, Heller S; NIHR DAFNE Research Study Group. The 5x1 DAFNE study protocol: a cluster randomised trial comparing a standard 5 day DAFNE course delivered over 1 week against DAFNE training delivered over 1 day a week for 5 consecutive weeks. BMC Endocr Disord. 2012 Nov 8;12:28. doi: 10.1186/1472-6823-12-28. PMID 23136929